CLINICAL TRIAL: NCT01719783
Title: Reactogenicity, Safety and Immunogenicity of a Live Monovalent A/17/Turkey/Turkey/05/133 (H5N2) Influenza Vaccine
Brief Title: Reactogenicity, Safety, and Immunogenicity of a Live Monovalent H5N2 Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Microgen (Other); Institute of Experimental Medicine, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAIV-H5N2-01
Record Dates: First submitted 2012-10-26; First posted 2012-11-01 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Influenza
Keywords: influenza; vaccine; pandemic
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAIV H5N2 (Experimental): Two doses of live monovalent influenza vaccine A/17/turkey/Turkey/05/133 ( live monovalent (LAIV H5N2) given intranasally
  Interventions: Biological: LAIV H5N2
- Placebo (Placebo Comparator): two doses of placebo solution intranasal
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: LAIV H5N2 — 2 doses provided intranasally
  Other Names: A/17/turkey/Turkey/05/133(H5N2)live influenza vaccine
  Arms: LAIV H5N2
Other: Placebo — 2 doses of placebo provided intranasally
  Arms: Placebo

SUMMARY:
To evaluate the safety profile of two intranasal doses of LAIV A/17/turkey/Turkey/05/133 (H5N2) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Legal male or female adult 18 through 49 years of age at the enrollment visit.
* Literate and willing to provide written informed consent.
* Free of obvious health problems, as established by the medical history and screening evaluations, including physical examination.
* Capable and willing to complete diary cards and willing to return for all follow-up visits
* Willing to comply with the rules of the isolation unit (including willing and able to take oseltamivir influenza antiviral medication, should that be recommended by a study physician).
* For females, willing to take reliable birth control measures throughout the entire period of participation in the study.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until four weeks after study completion.
* Practice of nasal irrigation on a regular basis within the past six months or has engaged in nasal irrigation within two weeks prior to enrollment.
* Recent history of frequent nose bleeds (>5 within the past year).
* Clinically relevant abnormal paranasal anatomy.
* Recent history (within the past month) of rhino or sinus surgery, or surgery for any traumatic injury of the nose.
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Other acute illness at the time of study enrollment.
* Receipt of immune globulin or other blood products within three months prior to study enrollment or planned receipt of such products during the period of subject participation in the study.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, 0.5 mg per kg per day; topical steroids are allowed, exclusive of nasal.)
* Participation in any previous trial of any H5 or H7 containing influenza vaccine.
* History of asthma.
* Hypersensitivity after previous administration of any influenza vaccine.
* History of wheezing after past receipt of any live influenza vaccine.
* Other adverse event (AE) following immunization, at least possibly related to previous receipt of any influenza vaccine.
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein.
* Seasonal (autumnal) hypersensitivity to the natural environment.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, metabolic, neurologic, psychiatric or renal functional abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives. Subjects with physical examination findings or clinical laboratory screening results which would be graded 2 or higher on the AE severity grading scale (see Attachments) will be excluded from entry into the study and will be excluded from receipt of dose two of study vaccine or placebo.
* History of leukemia or any other blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressive or immunodeficient condition of any kind, including HIV infection.
* Known chronic hepatitis B (HBV) or hepatitis C (HCV) infection.
* Known tuberculosis infection or evidence of previous tuberculosis exposure.
* History of chronic alcohol abuse and/or illegal drug use.
* Claustrophobia or sociophobia.
* Pregnancy or lactation. (A negative pregnancy test will be required before administration of study vaccine or placebo for all women of childbearing potential.)
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if he/she participates in the study or would interfere with the evaluation of the study objectives

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Influenza, Saint Petersburg, Russia

REFERENCES:
- [Derived] Kiseleva I, Dubrovina I, Fedorova E, Larionova N, Isakova-Sivak I, Bazhenova E, Pisareva M, Kuznetsova V, Flores J, Rudenko L. Genetic stability of live attenuated vaccines against potentially pandemic influenza viruses. Vaccine. 2015 Dec 8;33(49):7008-14. doi: 10.1016/j.vaccine.2015.09.050. Epub 2015 Oct 2. PMID 26432909
- [Derived] Rudenko L, Kiseleva I, Stukova M, Erofeeva M, Naykhin A, Donina S, Larionova N, Pisareva M, Krivitskaya V, Flores J; Russian LAIV Trial Study Group. Clinical testing of pre-pandemic live attenuated A/H5N2 influenza candidate vaccine in adult volunteers: results from a placebo-controlled, randomized double-blind phase I study. Vaccine. 2015 Sep 22;33(39):5110-7. doi: 10.1016/j.vaccine.2015.08.019. Epub 2015 Aug 19. PMID 26296497

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: two doses of placebo solution provided intranasally
Period: Dose 1
Arm/Group | LAIV H5N2 | Placebo
Started | 30 | 10
Completed | 30 | 10
Not Completed | 0 | 0
Period: Dose 2
Arm/Group | LAIV H5N2 | Placebo
Started | 30 | 10
Completed | 29 | 10
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAIV H5N2 | Placebo | Total
Number analyzed (Participants) | 30 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (10.4) | 29.2 (10.8) | 28.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 21 | 6 | 27
Region of Enrollment [Number; unit: participants]
  Russia | 30 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events by Severity
Description: Occurrence of participants with adverse events associated with intranasal administration, by worst grade of severity
Time Frame: 6 days
Population: All participants that received either a vaccine or placebo, by dose
Measure: Count of Participants; unit: Participants
Groups:
- Dose 1: Vaccine: Received dose 1 of vaccine
- Dose 1: Placebo: Received Dose 1 of Placebo
- Dose 2: Vaccine: Received Dose 2 of vaccine
- Dose 2: Placebo: Received Dose 2 of placebo
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Worst grade: mild | 20 | 8 | 25 | 8
  Worst grade: moderate | 1 | 0 | 0 | 0
  Worst grade: severe | 0 | 0 | 0 | 0
  None | 9 | 2 | 4 | 2

2. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for Serum Hemagglutination Inhibition (HAI)
Description: Defined as a four-fold or greater antibody rise in titer from pre-vaccination level.
  HAI = hemagglutination-inhibition, conducted using World Health Organization (WHO)-recommended protocols.
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Participants receiving study vaccine or placebo and with pre- and post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Seroconversion | 4 | 0 | 11 | 0
  No seroconversion | 26 | 10 | 18 | 10

3. Secondary Outcome: Number/Percentage of Subjects With Serum Neutralizing Antibodies
Description: Defined as a four-fold or greater antibody rise in titer from pre-vaccination level.
  Measured by microneutralization assay in Madin-Darby canine kidney cells (MDCK).
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Participants receiving study vaccine or placebo and with pre- and post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Seroconversion | 3 | 0 | 14 | 0
  No seroconversion | 27 | 10 | 15 | 10

4. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for Serum Immunoglobulin A (IgA)
Description: IgA = immunoglobulin class A antibodies Determined using ELISA using whole purified H5N2
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Participants receiving study vaccine or placebo and with pre- and post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Seroconversion | 0 | 0 | 2 | 0
  No seroconversion | 30 | 10 | 27 | 10

5. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for Serum Immunoglobulin G (IgG)
Description: Determined using ELISA using whole purified H5N2.
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Participants receiving study vaccine or placebo and with pre- and post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Seroconversion | 0 | 0 | 1 | 0
  No seroconversion | 30 | 10 | 28 | 10

6. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for Secretory IgA
Description: IgA antibodies from the nasal mucosa detected in nasal wick specimens. Determined using ELISA using whole purified H5N2
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Participants receiving study vaccine or placebo and with pre- and post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Seroconversion | 2 | 0 | 6 | 0
  No seroconversion | 28 | 10 | 23 | 10

7. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for IgA in Saliva
Description: IgA = Immunoglobulin Class A antibodies. Determined using ELISA using whole purified H5N2.
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Participants receiving study vaccine or placebo and with pre- and post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Seroconversion | 3 | 0 | 10 | 0
  No seroconversion | 27 | 10 | 19 | 10

8. Secondary Outcome: Number/Percentage of Vaccinated Participants Shedding Influenza Virus After First Dose
Description: Nasal swabs were collected and used for Reverse transcription polymerase chain reaction (rRTPCR) assays to detect shedding of influenza virus for days 1-6 of the study.
Time Frame: 6 days post-vaccination
Population: Participants receiving first dose of study vaccine and with post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Groups:
- Day 1: Shedding 1 day after first dose was administered
- Day 2: Shedding 2 days after first dose was administered
- Day 3: Shedding 3 days after dose was administered
- Day 4: Shedding 4 days after dose was administered
- Day 5: Shedding 5 days after dose was administered
- Day 6: Shedding 6 days after dose was administered
Arm/Group | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 30
Participants
  Shedding | 28 | 5 | 0 | 0 | 0 | 0
  No shedding | 2 | 25 | 30 | 30 | 30 | 30

9. Secondary Outcome: Number/Percentage of Vaccinated Participants Shedding Influenza Virus After Second Dose
Description: Nasal swabs were collected and used for Reverse transcription polymerase chain reaction (rRTPCR) assays to detect shedding of influenza virus for days 29-34 of the study (6 days after the second vaccination).
Time Frame: 6 days post-vaccination
Population: Participants receiving second dose of study vaccine and with post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Arm/Group | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29 | 29
Participants
  Shedding | 21 | 4 | 0 | 0 | 0 | 0
  No shedding | 8 | 25 | 29 | 29 | 29 | 29

10. Secondary Outcome: Geometric Mean Titers for Serum HAI Antibodies
Description: Geometric mean titers for serum hemagglutination inhibition antibodies
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: Participants receiving both doses of study vaccine or placebo and with pre- and post-vaccination immunologic parameters measured
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | LAIV H5N2 | Placebo
Number analyzed (Participants) | 29 | 10
titer
  Day 0 | 2.5 [2.5 to 2.5] | 2.7 [2.3 to 3.1]
  After dose 1 | 3.5 [2.9 to 4.2] | 2.7 [2.3 to 3.1]
  After dose 2 | 4.7 [3.6 to 6.1] | 2.9 [2.1 to 3.9]

11. Secondary Outcome: Geometric Mean Titers (GMT) for Serum Neutralizing Antibodies
Description: Geometric mean titers for serum neutralizing antibodies measured by microneutralization assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | LAIV H5N2 | Placebo
Number analyzed (Participants) | 29 | 10
titer
  Day 0 | 5.2 [4.9 to 5.6] | 5.4 [4.6 to 6.3]
  After dose 1 | 6.7 [5.6 to 8.0] | 5.4 [4.6 to 6.3]
  After dose 2 | 11.8 [8.7 to 16] | 5.7 [4.7 to 7.1]

12. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD8+ IFNγ+ Responses
Description: Nasal swabs from days 1, 2, 3, 5, and 7 after the first vaccination and on days 1 and 3, corresponding to days 29 and 31,respectively, after the second dose were tested for viral shedding by inoculation in 10- to 11-day-old embryonated chicken eggs (ECE) followed by incubation at 32◦C for 72 h. Influenza virus was detected by standard hemagglutination test with 1% chicken red blood cells.
  An increase in the number of antigenic-specific T cells greater than 3 standard deviations over the mean placebo values was regarded as a positive T cell response.
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Participants receiving study vaccine or placebo and with pre- and post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Groups:
- Dose 1 or 2: Vaccine: Received dose 1 or 2 of vaccine
- Dose 1 or 2: Placebo: Received dose 1 or 2 of placebo
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo | Dose 1 or 2: Vaccine | Dose 1 or 2: Placebo
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 1 | 0 | 2 | 0 | 3 | 0
  No response | 28 | 10 | 27 | 10 | 26 | 10

13. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD4+ IFNγ+ Responses
Description: Nasal swabs from days 1, 2, 3, 5, and 7 after the first vaccination and on days 1 and 3, corresponding to days 29 and 31,respectively, after the second dose were tested for viral shedding by inoculation in 10- to 11-day-old ECE followed by incubation at 32◦C for 72 h. Influenza virus was detected by standard hemagglutination test with 1% chicken red blood cells.
  An increase in the number of antigenic-specific T cells greater than 3 standard deviations over the mean placebo values was regarded as a positive T cell response.
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Participants receiving study vaccine or placebo and with pre- and post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Groups:
- Dose 1: Vaccine: After receiving dose 1 of vaccine
- Dose 1: Placebo: After receiving Dose 1 of Placebo
- Dose 2: Vaccine: After receiving Dose 2 of vaccine
- Dose 2: Placebo: After receiving Dose 2 of placebo
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo | Dose 1 or 2: Vaccine | Dose 1 or 2: Placebo
Number analyzed (Participants) | 29 | 10 | 30 | 10 | 29 | 10
Participants
  Positive response | 3 | 0 | 5 | 0 | 6 | 0
  No response | 26 | 10 | 25 | 10 | 23 | 10

14. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD8+ IFNγ+ Effector Memory T Cell Responses
Description: Nasal swabs from days 1, 2, 3, 5, and 7 after the first vaccination and on days 1 and 3, corresponding to days 29 and 31,respectively, after the second dose were tested for viral shedding by inoculation in 10- to 11-day-old ECE followed by incubation at 32◦C for 72 h. Influenza virus was detected by standard hemagglutination test with 1% chicken red blood cells.
  An increase in the number of antigenic-specific T cells greater than 3SD over the mean placebo values was regarded as a positive T cell response.
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo | Dose 1 or 2: Vaccine | Dose 1 or 2: Placebo
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 6 | 0 | 3 | 0 | 8 | 0
  No response | 23 | 10 | 26 | 10 | 21 | 10

15. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD4+ IFNγ+ Central Memory T Cell Responses
Description: as for outcome 14
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo | Dose 1 or 2: Vaccine | Dose 1 or 2: Placebo
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 5 | 0 | 6 | 0 | 8 | 0
  No response | 24 | 10 | 23 | 10 | 21 | 10

16. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD4+ IFNγ+ Effector Memory T Cell Responses
Description: as for outcome 14
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Groups:
- Dose 1 or 2: Vaccine: After receiving dose 1 or 2 of vaccine
- Dose 1 or 2: Placebo: After receiving dose 1 or 2 of placebo
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo | Dose 1 or 2: Vaccine | Dose 1 or 2: Placebo
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 5 | 0 | 6 | 0 | 11 | 0
  No response | 24 | 10 | 23 | 10 | 18 | 10

17. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD8+ IFNγ+ Central Memory T Cell Responses
Description: as for outcome 14
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo | Dose 1 or 2: Vaccine | Dose 1 or 2: Placebo
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 2 | 1 | 6 | 3 | 3 | 0
  No response | 27 | 9 | 23 | 7 | 26 | 10

ADVERSE EVENTS:
Time Frame: Within 7 days of administration of dose
Description: Definition of adverse event does not differ from clinicaltrials.gov.
  Adverse events occurring during the 6 days following any dose, measured as observed by study staff or reported by the subject to study staff. This includes abnormal laboratory findings from blood and urine specimens collected on Days 6 and 34.
Arm/Group | Dose 1: Vaccine | Dose 1: Placebo | Dose 2: Vaccine | Dose 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/10 | 0/29 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/10 | 0/29 | 0/10
Other Adverse Events (participants affected / at risk) | 21/30 | 8/30 | 25/30 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1: Vaccine (N=30) | Dose 1: Placebo (N=30) | Dose 2: Vaccine (N=30) | Dose 2: Placebo (N=10)
Alanine Aminotransferase Increased (Investigations) | 1 | 1 | 3 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 1 | 1 | 0
Blood Alkaline Phopsphatase Decreased (Investigations) | 1 | 0 | 0 | 1
Blood Bicarbonate Increased (Investigations) | 14 | 7 | 15 | 4
Blood Bilirubin Increased (Investigations) | 1 | 0 | 3 | 0
Blood Calcium Increased (Investigations) | 5 | 1 | 4 | 1
Blood Potassium Increased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin Increased (Investigations) | 3 | 2 | 7 | 2
Lymphocyte Count Increased (Investigations) | 1 | 0 | 10 | 3
Monocyte Count Increased (Investigations) | 1 | 0 | 3 | 1
Red Blood Cell Count Decreased (Investigations) | 1 | 0 | 3 | 0
White Blood Cell Count Increased (Investigations) | 1 | 0 | 2 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 6 | 1
Haematocrit Decreased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 4 | 2
Mean Cell Haemoglobin Concentraion Increased (Investigations) | 0 | 0 | 2 | 0
Mean Cell Volume Decreased (Investigations) | 0 | 0 | 1 | 0
Mean Platelet Volume Decreased (Investigations) | 0 | 0 | 1 | 0
Protein Total Increased (Investigations) | 0 | 0 | 1 | 0
Red Blood Cell Sedimentation Decreased (Investigations) | 0 | 0 | 2 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 3 | 5

LIMITATIONS AND CAVEATS:
Study was completed as expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No